CLINICAL TRIAL: NCT01479686
Title: 3.0T High-field Intraoperative MRI Guided Extent of Resection in Cerebral Glioma Surgery: a Single Center Prospective Randomized Triple-blind Controlled Clinical Trial
Brief Title: iMRI Guided Resection in Cerebral Glioma Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jinsong Wu, M.D.,Ph.D., Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XBR2011022
Record Dates: First submitted 2011-11-19; First posted 2011-11-24 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Glioma
Keywords: GLIOMA; NEURONAVIGATION; INTERVENTIONAL MRI
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional neuronavigation (Active Comparator): conventional neuronavigation guided resection in adults with glioma
  Interventions: Procedure: conventional neuronavigation
- intraoperative MRI (Experimental): iMRI guided resection in adults with glioma
  Interventions: Procedure: iMRI

INTERVENTIONS:
Procedure: iMRI — 3.0TiMRI guided resection in adults with glioma
  Arms: intraoperative MRI
Procedure: conventional neuronavigation — conventional neuronavigation guided resection in adults with glioma
  Arms: conventional neuronavigation

SUMMARY:
Many clinical studies have been reported on iMRI, however, their evidence levels are relatively not as good as what people hope they will be. Based on the available literature, there is, at best, level 2 evidence that iMRI-guided surgery is more effective than conventional neuronavigation-guided surgery.

The investigators aim to do a single center prospective randomized triple-blind controlled clinical trial to assess the effect of 3.0T high-field intraoperative MRI-guided glioma resection on surgical efficiency and progression-free survival of malignant glioma to provide a level 2A evidence for its clinical application.

DETAILED DESCRIPTION:
Since the first introduction of the GE Signa System by the Brigham and Women's Hospital as the world's first intraoperative MRI in 1993, iMRI has been so increasingly applied that it has been one of the most important techniques and concepts in the field of neurosurgery. Many clinical studies have been reported on this respect, however, their evidence levels are relatively not as good as what people hope they will be.Based on the available literature, there is, at best, level 2B evidence that iMRI-guided surgery is more effective than conventional neuronavigation-guided surgery.

Rationale: Intraoperative magnetic resonance imaging (MRI)-guided intracranial surgery, one of whose most frequently reported indications is cerebral glioma surgery, may help update images for navigational systems, providing data on the extent of resection and localization of tumor remnants, and thereby enable intraoperative reliable immediate resection control to eliminate the effect of brain shift on the extent of resection. Intraoperative MRI systems can be divided into low-field intraoperative MRI(0.5T or less) and high-field intraoperative MRI (1.5T or more) according to their various field strengths. The latter enables intraoperative imaging at higher quality and more available imaging modalities but with more cost and equipment requirements.

Purpose: We aim to do a single center prospective randomized triple-blind controlled clinical trial to assess the effect of 3.0T high-field intraoperative MRI-guided glioma resection on surgical efficiency and progression-free survival of malignant glioma. We hypothesize that the use of high-field intraoperative MRI will enable more complete tumor resection than conventional neuronavigation-guided resection,reducing the morbidity and leading to more improved progression-free survival and quality of life in patients with malignant glioma.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18-70 years with highly suspected (as assessed by study surgeon), newly diagnosed, untreated malignant glioma (see appendix 1)
2. Individuals with supratentorial gliomas with bodies involving in frontal lobe, temporal lobe, parietal lobe, occipital lobe or insular lobe
3. Individuals with the preoperative assessment that radiological radicality should be achieved
4. Individuals either with or without tumor in eloquent areas (see appendix 2)
5. Karnofsky performance scale 70 or more
6. All patients gave written informed consent.

Appendix 1. Histological types（WHO 2007）:

1. Astrocytic tumours:Pilomyxoid astrocytoma 9425/3 Pleomorphic xanthoastrocytoma 9424/3 Diffuse astrocytoma 9400/3 Fibrillary astrocytoma 9420/3 Gemistocytic astrocytoma 9411/3 Protoplasmic astrocytoma 9410/3 Anaplastic astrocytoma 9401/3 Glioblastoma 9440/3 Giant cell glioblastoma 9441/3 Gliosarcoma 9442/3
2. Oligodendroglial tumours:Oligodendroglioma 9450/3 Anaplastic oligodendroglioma 9451/3
3. Oligoastrocytic tumours:Oligoastrocytoma 9382/3 Anaplastic oligoastrocytoma 9382/3
4. Ependymal tumours:Ependymoma 9391/3 Cellular 9391/3 Papillary 9393/3 Clear cell 9391/3 Tanycytic 9391/3 Anaplastic ependymoma 9392/3

Morphology code of the International Classification of Diseases for Oncology (ICD-O) {614A} and the Systematized Nomenclature of Medicine (http://snomen.org). Behaviour is coded /0 for benign tumours, /3 for malignant tumours and /1 for borderline or uncertain behaviour.

Tumor grade: grade II~IV according to the latest WHO grading criteria;

Appendix 2. Tumor location in eloquent areas:

located in or close to areas of the dominant-hemisphere that associated with motor or language functions, including:

1. Frontal lobe, which divided into inferior frontal gyrus (BA44-Pars opercularis, BA45-Pars triangularis/Broca's area), middle frontal gyrus (BA9, BA46), superior frontal gyrus (BA4, BA6, BA8), primary motor cortex (BA4), premotor cortex (BA6), and supplementary motor area (BA6)
2. Parietal lobe, which divided into inferior parietal lobule (BA40-supramarginal gyrus, BA39-angular gyrus), parietal operculum (BA43), and primary somatosensory cortex (BA1, BA2, BA3)
3. Temporal lobe, which divided into transverse temporal gyrus (BA41, BA42), superior temporal gyrus (BA38, BA22/Wernicke's area), middle temporal gyrus (BA21)
4. Insular lobe.

Exclusion Criteria:

1. Individuals with age < 18 years or > 70 years
2. Tumours of the midline, basal ganglia, cerebellum, or brain stem
3. Recurrent gliomas after surgery (except needle biopsy)
4. Primary gliomas with history of radiotherapy or chemotherapy
5. Contraindications precluding intraoperative MRI-guided surgery
6. Inability to give informed consent
7. KPS < 70
8. Renal insufficiency or hepatic insufficiency
9. History of malignant tumours at any body site
10. Tumour locations (in important eloquent area) do not enable complete resection of tumour.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2011-09; Primary Completion 2018-09 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Extent of resection | 3 years
  Extent of resection (EOR) based on early postoperative MRI obtained within 72 h after surgery. Gross total resection (GTR) was defined as the complete disappearance of all enhancing lesions (T1WI) for HGG and the complete disappearance of all nonenhancing (T2WI FLAIR) lesions for LGG. The EOR were quantitatively volumetric analyses for all gliomas and gliomas grouped according to eloquent areas and non-eloquent areas, and stratified as: GTR, 100% resection; subtotal resection ≥ 90% resection, partial resection ≥ 70% resection, biopsy, resection ≥98% for OS advantage (HGG) and resection ≥90% for OS advantage (LGG).

SECONDARY OUTCOMES:
OS | 10 years
  Overall survival analyses for all gliomas and gliomas grouped according to eloquent areas and non-eloquent areas.
PFS | 10 years
  Neuropathological confirmed non-glioma lesions or benign histologies are excluded from the secondary endpoints follow up. All participants were observed, with serial clinical evaluations and MRI scans every 3 months following interventions, which was the routine for these diseases. Progression was deﬁned in accordance with RANO criteria.
Postoperative complications | after surgery
  Postoperative complications: e.g., postoperative epilepsy, infection, bleeding and infarction.
Health economics | after surgery
  Health economics: surgical time, surgical cost, postoperative hospitalization days, and hospitalization expenses
MRI-related adverse events | after surgery
  MRI-related adverse events: risks of airway management, burn, MRI mechanical damage, and other safety analysis.
Surgery related morbidity | 3 years
  Assessment of motor and language functions (Morbidity): whether there are newly postoperative hemiplegia or aphasia.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-fu Zhou, M.D., Study Chair — Huashan Hospital; Ying Mao, M.D., Ph.D, Principal Investigator — Huashan Hospital; Jin-song Wu, M.D., Ph.D, Principal Investigator — Huashan Hospital
Locations (1):
- Department of Neurologic Surgery, Huashan Hospital, Shanghai Medical College, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Fountain DM, Bryant A, Barone DG, Waqar M, Hart MG, Bulbeck H, Kernohan A, Watts C, Jenkinson MD. Intraoperative imaging technology to maximise extent of resection for glioma: a network meta-analysis. Cochrane Database Syst Rev. 2021 Jan 4;1(1):CD013630. doi: 10.1002/14651858.CD013630.pub2. PMID 33428222